CLINICAL TRIAL: NCT02475486
Title: Role of the Sympathetic Nervous System (ANS) Dysregulation in the Persistence of Fatigue in Rheumatoid Arthritis Patients Treated With Anti-TNF (Tumor Necrosis Factor) - a Monocentric Cross-sectional Study
Brief Title: Role of the ANS Dysregulation in the Persistence of Fatigue in Rheumatoid Arthritis Patients Treated With Anti-TNF
Acronym: ANSRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1508054; 2015-A00655-44 (Other: ANSM)
Record Dates: First submitted 2015-06-16; First posted 2015-06-18 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; sympathetic nervous system; SNA; fatigue
MeSH Terms: conditions — Arthritis, Rheumatoid; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high fatigue (Other): Measure of ANS by VistaO2 device in Rheumatoid arthritis (RA) patients with low disease activity according to DAS28 <3.2 with visual analog scale of fatigue is > 5
  Interventions: Device: VistaO2
- low fatigue (Other): Measure of ANS by VistaO2 device in Rheumatoid arthritis (RA) patients with low disease activity according to DAS28 <3.2 with visual analog scale of fatigue is < or equal to 5
  Interventions: Device: VistaO2

INTERVENTIONS:
Device: VistaO2 — ANS (sympathetic nervous system) parameters are measured by VistaO2 device in RA patients

SUMMARY:
Despite the large therapeutic arsenal available since one decade allowing a strong reduction of inflammation process, rheumatoid arthritis (RA) patients claimed pain, fatigue, sleep problems and other quality of life outcomes. Fatigue reduction during TNF blockers therapy is lower than the strong reduction in RA disease activity. Furthermore, RA patients have higher prevalence of non-inflammatory pain than general population. Fatigue is a real major problem due to 50% of patients considered it as severe.

This dissociation between disease activity and fatigue level suggests that fatigue is multifactorial. No consistent explanations for fatigue are currently available.

ELIGIBILITY:
Inclusion Criteria :

* RA diagnosis according to ACR/EULAR 2010
* RA with low disease activity according to DAS28 < 3.2
* Written consent obtained

Exclusion Criteria :

* Other diagnosis than RA
* Depression known
* Hypertension treated or not,
* Diseases interfering with ANS analysis: cardiac arrhythmia, beta-blocker therapy,
* Pregnant or breastfeeding women,
* Inability to go two consecutive days at the North hospital for the delivery and return of the Vista02 device

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Ratio low/high frequencies of power spectral density of R-R intervals | day1
  Comparison of Ratio low/high frequencies of power spectral density of R-R intervals between RA patients with low fatigue and RA patients with high fatigue. Ratio low/high frequencies of power spectral density of R-R is measured by VistaO2 device.

SECONDARY OUTCOMES:
Number of sleep apnea syndrome | day 1
  Comparison of Number of sleep apnea syndrome between between RA patients with low fatigue and RA patients with high fatigue. sleep apnea syndrome is measured by VistaO2 device.
Standard deviation of all R-R intervals (SDNN) | day 1
  Comparison of Standard deviation of all R-R intervals (SDNN) between RA patients with low fatigue and RA patients with high fatigue. Standard deviation of all R-R intervals (SDNN) is measured by VistaO2 device.
Total Power spectral density (PSD) | day 1
  Comparison of Total Power spectral density (PSD) between RA patients with low fatigue and RA patients with high fatigue. Total Power spectral density (PSD) is measured by VistaO2 device.
PSD of Lower Frequencies | day 1
  Comparison of PSD of Lower Frequencies between RA patients with low fatigue and RA patients with high fatigue. PSD of Lower Frequencies is measured by VistaO2 device.
PSD of High Frequencies | day 1
  Comparison of PSD of High Frequencies between RA patients with low fatigue and RA patients with high fatigue. PSD of High Frequencies is measured by VistaO2 device.
normalized value of the High and Low frequencies | day 1
  Comparison of normalized value of the High and Low frequencies between RA patients with low fatigue and RA patients with high fatigue. normalized value of the High and Low frequencies is measured by VistaO2 device.
Physical activity | day 1
  Comparison of physical activity between RA patients with low fatigue and RA patients with high fatigue. Physical activity is measured by IPAQ score.
quality of sleep | day 1
  Comparison of quality of sleep between RA patients with low fatigue and RA patients with high fatigue. Quality of sleep is measured by PSQI score.
depression | day 1
  Comparison of depression level between RA patients with low fatigue and RA patients with high fatigue. Depression is measured by HAD, BDI and HDRS scales.
Correlation between fatigue and Ratio low/high frequencies of power spectral density of R-R intervals | day 1
  fatigue is measured with a visual analogic scale

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Marotte, PUPH, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No